CLINICAL TRIAL: NCT02544477
Title: High-flow Nasal Cannula Oxygen Versus Conventional Oxygen Therapy After Pulmonary Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Maria Teresa Congedo, Medical Doctor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFNC after pulmonary lobectomy
Record Dates: First submitted 2015-08-26; First posted 2015-09-09 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Respiratory Insufficiency; Lung Cancer
MeSH Terms: conditions — Respiratory Insufficiency; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-flow nasal cannula oxygen (HFNCO) (Experimental): Patients will receive HFNCO treatment with a gas flow level = 50 L/min and a FiO2 set to maintain peripheral oxygen saturation (SpO2) of 92% - 98%.
  Interventions: Device: High-flow Nasal Cannula Oxygen (HFNCO)
- standard oxygen therapy (Active Comparator): Patients will receive oxygen treatment by means of a conventional face mask, with a level of fraction of inspired oxygen (FiO2) set to maintain peripheral oxygen saturation (SpO2) of 92% - 98%.
  Interventions: Device: Conventional oxygen treatment

INTERVENTIONS:
Device: High-flow Nasal Cannula Oxygen (HFNCO)
  Arms: High-flow nasal cannula oxygen (HFNCO)
Device: Conventional oxygen treatment
  Arms: standard oxygen therapy

SUMMARY:
The primary objective of this study is to evaluate the effect of early application of nasal high flow oxygen therapy after pulmonary lobectomy on the incidence of postoperative hypoxemia

DETAILED DESCRIPTION:
High-flow nasal cannula oxygen (HFNCO) treatment has been showed to have several clinical advantages compared with conventional oxygen therapy. Currently, no reports have described the effects of HFNCO in postoperative patients after thoracic surgery. The primary objective of this study is to determine the incidence of postoperative hypoxemia (defined as a PaO2/FiO2 ratio <300) in patients with lung cancer after pulmonary lobectomy.

In the postoperative period after extubation, patients will be randomly assigned to either:

1. standard oxygen therapy group (control group) or
2. HFNCO group (study group).

In the control group, patients will receive oxygen treatment by means of a conventional face mask, with a level of fraction of inspired oxygen (FiO2) set to maintain peripheral oxygen saturation (SpO2) = 92% - 98%. Patients in the study group will be given HFNCO treatment with a gas flow level = 50 L/min and a FiO2 set to maintain peripheral oxygen saturation (SpO2) = 92% - 98%. After 48 hours from study entry, all patients will be evaluated for possible interruption of oxygen treatment on the basis of their clinical conditions.

ELIGIBILITY:
Inclusion Criteria:

* planned pulmonary lobectomy for lung cancer

Exclusion Criteria:

* age <18 years
* patient refusal
* body mass index ≥35 kg/m2
* sleep apnea syndrome
* tracheostomy
* home oxygen therapy
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with hypoxemia (defined as a PaO2/FiO2 ratio <300) after pulmonary lobectomy in patients with lung cancer | during the first 96 hours after surgery

SECONDARY OUTCOMES:
Number of patients with SpO2 <93% in room air | after 48 hours from surgery and until 7th post operative day
Number of patients undergoing endotracheal intubation or non-invasive ventilation for acute respiratory failure | during the first 7 days after surgery
  Respiratory failure will be defined as the presence of at least two of the following:
  * respiratory acidosis (arterial pH ≤7.35 with PaCO2 ≥ 45 mm Hg);
  * SpO2 < 90% or PaO2 < 60 mmHg at an FiO2 ≥ 0.5;
  * respiratory frequency > 35/min;
  * altered state of consciousness;
  * clinical signs of respiratory muscle fatigue.
  Respiratory failure will be treated using noninvasive ventilation (NIV), except when endotracheal intubation (ETI) will be required, i.e., when any of the following clinical events will be present:
  * respiratory or cardiac arrest;
  * respiratory pauses with loss of consciousness or gasping;
  * psychomotor agitation inadequately controlled by sedation;
  * massive aspiration;
  * persistent inability to remove respiratory secretions;
  * heart rate < 50/min with loss of alertness;
  * severe hemodynamic instability without response to fluids and vasoactive drugs. Patients with deterioration of blood gases or tachypnea despite 1 hour of NIV will undergo ETI.
Postoperative pulmonary complications | during the first 7 days after surgery
Respiratory discomfort evaluated by VAS (visual analogic scale) ranging from 0 (no discomfort) to 10 (maximum imaginable discomfort) | during the first 96 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy

REFERENCES:
- [Derived] Pennisi MA, Bello G, Congedo MT, Montini L, Nachira D, Ferretti GM, Meacci E, Gualtieri E, De Pascale G, Grieco DL, Margaritora S, Antonelli M. Early nasal high-flow versus Venturi mask oxygen therapy after lung resection: a randomized trial. Crit Care. 2019 Feb 28;23(1):68. doi: 10.1186/s13054-019-2361-5. PMID 30819227